CLINICAL TRIAL: NCT04979143
Title: Moses Vaporization: Is Use of Moses 2.0 in Holmium Laser Ablation of the Prostate More Efficient
Acronym: Moses 2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment due to new alternative surgical treatment options emerging and being requested by patients.
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Don Neff, MD, FACS, Associate Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GU-EN-MOSES 2.0
Record Dates: First submitted 2021-07-16; First posted 2021-07-28 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HoLVP with the use of Moses 2.0 technology (Other): HoLVP with the use of Moses 2.0 technology
  Interventions: Procedure: Surgical Approach
- HoLVP without the use of Moses 2.0 technology (Other): HoLVP without the use of Moses 2.0 technology
  Interventions: Procedure: Surgical Approach

INTERVENTIONS:
Procedure: Surgical Approach — The surgical laser used will be randomized. All lasers used during this trial are all FDA approved devices and used per routine clinical care.

SUMMARY:
To determine if use of Moses 2.0 results in improved ablation efficiency during holmium laser vaporization of the prostate. To determine if use of Moses 2.0 results in less char, improved visibility, and improved hemostasis in prostate vaporization.

DETAILED DESCRIPTION:
Patients will be evaluated preoperatively per standard of care in urology clinic. We will obtain American Urological Association Symptom Score (AUA-SS) and Quality of Life (QoL) assessment as well as post-void residual bladder scan (PVR), and prostate specific antigen (PSA). All of these assessments will be part of standard of care.

Based on the current coronavirus (COVID-19) pandemic and the changing health landscape with increased emphasis on telehealth, patient may be offered virtual appointments for aspects of the trial that do not require in-person evaluation or testing. These include but are not limited to inclusion/exclusion criteria evaluation, consent for trial participation, or survey completion.

Patients will be taken to the operating room per standard of care. They will be randomized to either Holmium Laser Vaporization of Prostate (HoLVP) with or without the use of Moses 2.0 technology. The surgeon and patient will both be blinded to the laser mode.

HoLVP will occur in standard fashion thereafter utilizing at 550-micron holmium Xpeeda side fire laser fiber at settings of 2 Joules, 50 Hertz. Moses 2.0 will be activated or not by operating room personnel based on patient's randomization status. Again, the surgeon and assistant will not be informed of the Moses status.

Intraoperative parameters will be recorded including total procedure time, total vaporization time, vaporization efficiency (g/min), and total energy used. Surgeons will evaluate tissue char, visibility, hemostasis, as well as select if they think Moses 2.0 was activated or not for the procedure.

Timeline for catheter removal will be per surgeon discretion with a general plan for removal in the post-anesthesia care unit with trial of void before discharge on day of surgery. If patient is discharged with a catheter in place, removal date will be determined per surgeon's discretion.

Patients will be seen in urology clinic for follow up per standard of care at 6 weeks, 3 months, and 12 months post operatively at which time we will obtain symptom questionnaires. A PVR will be obtained at 6 weeks. PSA will be measured at 3 months post operatively, to act as a surrogate marker for percentage of tissue vaporized since it can be compared to pre-operative PSA.

Outcomes from surgery will be assessed including changing in AUA-SS and QoL, and PVR. We will also evaluate for complications such as urethral stricture, bladder neck contracture, and need for re-operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Patients with bothersome lower urinary tract symptoms who opt for surgical management
* Prostate size 60g or less

Exclusion Criteria:

* Current use of anticoagulation or antiplatelet agent Aspirin 81 use is okay and can be continued through the study
* Bleeding diathesis
* AUA symptom score < 9
* Current urinary retention
* Known diagnosis of prostate cancer
* Known diagnosis of neurogenic bladder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males only. Study is looking at benign prostate hyperplasia and lower urinary tract symptoms. Females do not have prostates
Enrollment: 19 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome is vaporization efficiency, measured in g/min | 5 years
  The primary outcome is vaporization efficiency, measured in g/min. For the purposes of this study, we defined improvement as at least a 50% improvement in ablation efficiency, based on improvements in enucleation efficiency observed in a recent study . Furthermore, based on a previous study we made of Moses 1.0, the ablation efficiency of Moses 1.0 is 1.77 g/min with a standard deviation of 1.41 g/min.7 Differences in ablation efficiency will be tested via Welch's t-test.10 Therefore, we calculated the sample size based on an anticipated improvement of efficiency to at least 2.66 g/min. We further allowed for a somewhat higher standard deviation for Moses 2.0 at 2 g/min, as the variance tends to increase as the efficiency increases. This resulted in an anticipated standardized effect size of approximately 0.51 standard deviations (moderate effect). At a significance level of 0.05 and 80% power, this means we will need 62 subjects per arm in the study.

SECONDARY OUTCOMES:
Tissue char, visibility, and hemostasis will be evaluated by the surgeon performing the procedure and ranked on a 10-point scale | 5 years
  Tissue char, visibility, and hemostasis will be evaluated by the surgeon performing the procedure and ranked on a 10-point scale. For these outcomes, we do not have as much preliminary data, however, it is reasonable to assume a moderate effect size, as was observed in a study of Holmium Laser Enucleation of Prostate (HoLEP) We will test for differences in the secondary outcomes using a multivariate ANOVA. The sample size for the primary outcome will provide greater than 80% power for this test, using the O'Brien and Shieh algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Neff, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No